CLINICAL TRIAL: NCT03920839
Title: A Phase 1b Combination Study of INCMGA00012 Plus Chemotherapy in Participants With Advanced Solid Tumors (POD1UM-105)
Brief Title: INCMGA00012 Plus Chemotherapy in Participants With Advanced Solid Tumors (POD1UM-105)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: As of November 4, 2019 the study was halted prematurely and will not resume.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-105
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Advanced and/or Metastatic Solid Tumors; Stage IIIB Not Amenable to Curative Therapy to Stage IV Non-small Cell Lung Cancer; Advanced/Metastatic Unresectable Malignant Pleural Mesothelioma
Keywords: solid tumors; non-small cell lung cancer; malignant pleural mesothelioma; chemotherapy; programmed cell death protein 1 (PD-1) inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Gemcitabine; Cisplatin; Pemetrexed; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- INCMGA00012 + gemcitabine/cisplatin (Experimental)
  Interventions: Drug: Retifanlimab; Drug: Gemcitabine; Drug: Cisplatin
- INCMGA00012 + pemetrexed/cisplatin (Experimental)
  Interventions: Drug: Retifanlimab; Drug: Cisplatin; Drug: Pemetrexed
- INCMGA00012 + pemetrexed/carboplatin (Experimental)
  Interventions: Drug: Retifanlimab; Drug: Pemetrexed; Drug: Carboplatin
- INCMGA00012 + paclitaxel/carboplatin (Experimental)
  Interventions: Drug: Retifanlimab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Retifanlimab — INCMGA00012 administered intravenously every 3 weeks.
  Other Names: INCMGA00012
Drug: Gemcitabine — Gemcitabine administered intravenously on Days 1 and 8 of 21-day cycles.
  Arms: INCMGA00012 + gemcitabine/cisplatin
Drug: Cisplatin — Cisplatin administered intravenously on Day 1 of 21-day cycles.
  Arms: INCMGA00012 + gemcitabine/cisplatin; INCMGA00012 + pemetrexed/cisplatin
Drug: Pemetrexed — Pemetrexed administered intravenously on Day 1 of 21-day cycles.
  Arms: INCMGA00012 + pemetrexed/carboplatin; INCMGA00012 + pemetrexed/cisplatin
Drug: Carboplatin — Carboplatin AUC5 or AUC6 administered intravenously on Day 1 of 21-day cycles.
  Arms: INCMGA00012 + paclitaxel/carboplatin; INCMGA00012 + pemetrexed/carboplatin
Drug: Paclitaxel — Paclitaxel administered intravenously on Day 1 of 21-day cycles.
  Arms: INCMGA00012 + paclitaxel/carboplatin

SUMMARY:
The purpose of this study is to assess the safety and tolerability and to determine the recommended Phase 2 dose of INCMGA00012 in combination with common standard-of-care chemotherapy regimens in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced and/or metastatic solid tumors including the following: histologically or cytologically confirmed diagnosis of Stage IIIB not amenable to curative treatment or Stage IV non-small cell lung cancer (pemetrexed-platinum treatment groups must have nonsquamous histology type); and histologically or cytologically confirmed diagnosis of advanced/metastatic unresectable malignant pleural mesothelioma.
* No prior systemic treatment with the following exceptions: participants with a known sensitizing mutation (eg, BRAF, EGFR, ALK, or ROS1) should have had disease progression on or following an approved targeted tyrosine kinase inhibitor; and participants who received adjuvant or neoadjuvant chemotherapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months before the date of enrollment.
* Measurable or nonmeasurable tumor lesions per RECIST v1.1.
* Eastern Cooperative Oncology Group performance status 0 to 1.

Exclusion Criteria:

* Received prior treatment with checkpoint inhibitor agents (such as anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4).
* Had major surgery within 3 weeks before the first dose of study treatment.
* Received radiation therapy to the lung(s) that is > 30 Gy within 6 months of the first dose of study treatment.
* Received palliative radiotherapy within 7 days before the first dose of study treatment.
* Has ≥ Grade 2 residual toxicities from the most recent prior therapy (except alopecia).
* Organ function (renal, hepatic), bone marrow reserve, and coagulation panel outside the protocol-defined laboratory values.
* Is currently participating and receiving investigational therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks before the first dose of study treatment.
* Has active autoimmune disease requiring systemic immunosuppression with corticosteroids (> 10 mg once daily of prednisone or equivalent) or immunosuppressive drugs within 2 years before the first dose of study treatment.
* Is on chronic systemic steroids (> 10 mg once daily of prednisone or equivalent).
* Known active central nervous system metastases and/or carcinomatous meningitis (patients with previously-treated and clinically stable brain metastases are eligible and a washout period of ≥ 4 weeks since radiation therapy is required).
* Known additional malignancy that is progressing or requires active treatment.
* Evidence of interstitial lung disease or active, noninfectious pneumonitis.
* History of organ transplant, including allogeneic stem cell transplantation.
* Active infections requiring systemic antibiotics.
* Known active hepatitis B or C.
* Has a diagnosis of immunodeficiency, including participants known to be HIV positive (positive for HIV 1/2 antibodies).
* Significant cardiac event within 6 months before Cycle 1 Day 1.
* Has received a live vaccine within 28 days of the planned start of study treatment.
* Known hypersensitivity to any component of the study drugs, excipients, or another monoclonal antibody which cannot be controlled with standard measures (eg, antihistamines and corticosteroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events with INCMGA00012 in combination with chemotherapy | Up to approximately 27 months
  Adverse events reported for the first time or worsening of a pre-existing event after the first dose of study treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, up to approximately 31 months
  Defined as the percentage of participants having complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as determined by investigator assessment.
Duration of response (DOR) | Through study completion, up to approximately 31 months
  Defined as the time from an initial objective response (CR or PR) according to RECIST v1.1 until disease progression as determined by investigator assessment or death due to any cause.
Disease control rate (DCR) | Through study completion, up to approximately 31 months
  Defined as the number of participants with CR or PR as best response or stable disease that was maintained for at least 12 weeks.
Cmax of INCMGA00012 when given in combination with chemotherapy agents | Through post-induction Cycle 5 Day 1, up to 15 weeks
  Maximum observed plasma or serum concentration.
Tmax of INCMGA00012 when given in combination with chemotherapy agents | Through post-induction Cycle 5 Day 1, up to 15 weeks
  Time to maximum concentration.
Cmin of INCMGA00012 when given in combination with chemotherapy agents | Through post-induction Cycle 5 Day 1, up to 15 weeks
  Minimum observed plasma or serum concentration over the dose interval.
AUC0-t of INCMGA00012 when given in combination with chemotherapy agents | Through post-induction Cycle 5 Day 1, up to 15 weeks
  Area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation

IPD SHARING:
Plan to Share IPD: No